CLINICAL TRIAL: NCT00207077
Title: A Phase I Study of Cetuximab in Combination With Erlotinib in Patients With Advanced Solid Malignancies
Brief Title: Study of Cetuximab in Combination With Tarceva in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-101
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Cetuximab; Erlotinib Hydrochloride

ARMS (1):
- A (Experimental)
  Interventions: Drug: Cetuximab + Erlotinib

INTERVENTIONS:
Drug: Cetuximab + Erlotinib — IV solution + tablet, IV+ oral, ERB 100 mg/m2, 200 mg/m2, 250 mg/m2 IV + Erl 150 mg tablet, ERB weekly/ Erl once daily, Until disease progression.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to find a safe and effective dose of the combination of cetuximab (Erbitux) and Tarceva (erlotinib).

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease
* Life expectancy of at least 3 months
* Must have at least one prior chemotherapy containing a platinum

Exclusion Criteria:

* Known or documented brain metastases
* Prior cetuximab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of the combination of Tarceva and Erbitux

SECONDARY OUTCOMES:
Radiographic response

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States